CLINICAL TRIAL: NCT06868641
Title: The TAIL-PrEP Study: Acceptability and Feasibility of a Tailored Adherence Intervention for Safe Discontinuation of Long-acting PrEP
Brief Title: The TAIL-PrEP Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kathrine Meyers, Associate Professor of Bio-Behavioral Sciences, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAU7044; 1R21MH133755-01 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: HIV Prevention; PrEP; Cabotegravir; Long-Acting Injectable; Acceptability; Feasibility
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAIL-PrEP (Experimental): Patients receiving the TAIL-PrEP intervention
  Interventions: Behavioral: TAIL-PrEP

INTERVENTIONS:
Behavioral: TAIL-PrEP — The TAIL-PrEP intervention is comprised of two components: (1) monthly cab-LA monitoring with specimens self-collected by patient and mailed to a lab for processing; and (2) monthly HIV prevention coaching with personalized cab-LA feedback.

SUMMARY:
The goal of the TAIL-PrEP study is to understand how to support the safe discontinuation of injectable long-acting cabotegravir (cab-LA) while maximizing the public health impact of biomedical HIV prevention interventions. In Aim 1, the study will pilot test and assess the acceptability and feasibility of the TAIL-PrEP intervention, which will use cabotegravir drug level monitoring to provide personalized HIV prevention coaching to patients discontinuing long-acting cab-LA. In Aim 2, the study will refine the TAIL-PrEP intervention and implementation strategy based on findings from the pilot study.

DETAILED DESCRIPTION:
Oral PrEP is highly effective but underutilized, with only 25% of individuals eligible for PrEP in the US having a prescription. Recent approval of cabotegravir-LA (cab-LA), a long-acting injectable integrase inhibitor and the first long-acting injectable PrEP, presents an opportunity to increase uptake. However, the long and variable half-life of cab-LA across different individuals after discontinuation (called the "tail") poses an implementation challenge. During the tail, cabotegravir levels are sub-therapeutic but could select for integrase-inhibitor resistance if the patient were to acquire HIV. This concern about the tail presents a barrier to providers prescribing cab-LA, potentially limiting the contribution of cab-LA to achieving End the HIV Epidemic targets and PrEP uptake and HIV infection. Currently, to mitigate this risk, individuals are advised to use oral PrEP for up to and beyond 12 months after stopping cab-LA injections if they have an ongoing risk of becoming infected with HIV. However, a risk mitigation strategy that requires daily oral PrEP may not be feasible or acceptable to many patients who started injectable PrEP precisely because they were unable or unwilling to adhere to a daily medication. The goal of the TAIL-PrEP study is to pilot test and assess the acceptability and feasibility of the TAIL-PrEP intervention, which will use cabotegravir drug levels measured in blood specimens to provide personalized feedback and HIV prevention coaching (Aim 1); and refine the TAIL-PrEP intervention and implementation strategy based on findings from the pilot study (Aim 2).

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* Have discontinued cab-LA injections within the last three months
* Not currently on cab-LA injections
* HIV-negative (self-report)
* Able to speak and read in English or Spanish,
* Able to receive and send monthly packages
* Have access to an internet-connected device capable of running the Zoom video conferencing platform
* Have a private location at which to take Zoom calls

The study period will end for patient participants once the monthly blood draw result indicates that cab-LA levels are not detectable (estimated average of 6 months across all patients) or after 6 months of the study, whichever comes first. If at 6 months of study participation, cab-LA levels are still detectable and participants adhered to at least 50% of study activities (self-collecting and mailing monthly blood samples, completing monthly surveys, attending monthly coaching sessions), participants will be invited to participate in the study for an additional 6 months, for a total of up to 12 study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability among Patients | 6 months
  Acceptability of the intervention will be assessed using the validated Acceptability of Intervention Measure (AIM). AIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from 1="completely disagree" to 5="completely agree". The AIM is scored by averaging responses across the 4 items. A higher average score indicates greater acceptability, which is a better outcome.
Feasibility among Patients | 6 months
  Feasibility of the intervention will be assessed using the validated Feasibility of Intervention Measure (FIM). FIM is a 4-item scale where respondents rate each item using a 5-point ordinal scale that ranges from 1="completely disagree" to 5="completely agree". The FIM is scored by averaging responses across the 4 items. A higher average score indicates greater feasibility, which is a better outcome.

SECONDARY OUTCOMES:
Adherence to TAIL-PrEP intervention | 6 months
  Adherence to the intervention will be assessed by calculating the proportion of intervention components completed out of components possible.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine A Meyers, DrPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided